CLINICAL TRIAL: NCT06337903
Title: Self-compassion for People with Multiple Sclerosis: an Exploratory Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Simpson (Other)
Responsible Party: Sponsor-Investigator, Robert Simpson, Investigator, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Self-compassion for PwMS
Record Dates: First submitted 2024-03-19; First posted 2024-03-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis; Self-Compassion
Keywords: Mindfulness
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-compassion intervention (Experimental): 8-week manualized online Mindful Self-Compassion course
  Interventions: Behavioral: Self-compassion intervention (the Mindful Self-Compassion course)

INTERVENTIONS:
Behavioral: Self-compassion intervention (the Mindful Self-Compassion course) — An online 8-week mindful self-compassion course with weekly sessions.

SUMMARY:
The goal of this clinical trial is to develop and investigate a compassion-based intervention (Mindful Self-Compassion course) in people with multiple sclerosis. The main objectives are:

1. Explore feasibility of trial processes including recruitment, adherence, retention, and follow-up
2. Explore experiences of people with multiple sclerosis with the Compassion-based intervention, including perceived effects, barriers and facilitators to participation, suggestions for improvement
3. Determine potential effects on stress, anxiety, depression, emotion regulation, illness adjustment, and self-compassion.

Participants will be asked to take part in an 8-week online Mindful Self-Compassion course and report changes in levels of stress, anxiety, depression, self-compassion, adjustment, emotion, and quality of life from pre- to post-intervention and at 3-month follow-up. Additionally, participants will be asked to take part in a semi-structured interview to explore their experiences with the course, perceived effects, and suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Able to understand spoken and written English
3. Have a neurologist-confirmed diagnosis of multiple sclerosis
4. Willing to take place in an Mindful Self Compassion course

Exclusion Criteria:

1. Cognitive impairment (<26 on the Montreal Cognitive Assessment)
2. Severe active mental health impairment (psychosis, suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 4 months
  The investigators will measure the number of participants eligible for and recruited to the study.
Retention | 4 months
  The investigators will measure the percentage of participants who complete outcome data.
Adherence | 4 months
  The investigators will measure the number of participants who completed the mindful self-compassion course.
Follow-up rates | 4 months
  The investigators will measure the percentage of participants who complete outcome measures pre-intervention, post-intervention, and at 3 months post-intervention.

SECONDARY OUTCOMES:
Stress | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Perceived Stress Scale-10. The total score can range from 0-40, with higher scores indicating higher perceived stress.
Anxiety | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Hospital Anxiety and Depression Scale. The total score ranges from 0-21, with higher values representing increased anxiety symptoms.
Depression | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Hospital Anxiety and Depression Scale. The total score ranges from 0-21, with higher values representing increased depressive symptoms.
Self-compassion | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Self-Compassion Scale - Short Form. The total score ranges from a 1-5 Likert scale, with higher scores representing high self-compassion.
Emotion Regulation | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Difficulties in Emotion Regulation Scale - Short Form. Answers are assessed using a 5-point Likert scale. Higher values indicate greater difficulties in emotion regulation.
Quality of Life using the Multiple Sclerosis Impact Scale (MSIS-29) | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Multiple Sclerosis Impact Scale. Items on the scale have a Likert scale from 1-5, with a range of 0-100 total and higher scores indicating greater disability.
Participant Experiences and Perspectives | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Semi-structured interviews will aim to capture participants' experiences with the course and perspectives on the use of self-compassion in care.
Adjustment | Measured at baseline, 8-week follow-up, and 3-month follow-up.
  Measured using the Coping with MS Scale. Answers are assessed using a 5-point Likert scale and a mean per subscale group will be reported. Higher values indicate greater tendency to use coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simpson, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No